CLINICAL TRIAL: NCT03855852
Title: Evaluation Of Vertical Bone Gain Following One Stage Ridge Augmentation With Advanced Platelet Rich Fibrin (A-PRF) And Xenograft Compared to Guided Bone Regeneration Using Collagen Membrane and Xenograft.
Brief Title: Evaluation of Vertical Bone Gain After Ridge Augmentation With APRF & Xenograft Vs Collagen Membrane & Xenograft. RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdallah waleed sobhi Shbair, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-02-15
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Bone Loss, Alveolar
Keywords: vertical bone defect; Ridge augmentation; One stage; Xenograft; Collagen membrane; Advanced platelet rich fibrin; Guided bone regeneration; Surgical template; Implant; horizontal bone defect
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
  * A Randomized clinical trial
  * Parallel study group
  * A trial will be carried out in outpatient clinic of Periodontology Department ,Faculty of Dentistry , Cairo University .
  * Equal randomization with equal probabilities for intervention.
  * Positive controlled : Both groups will receive treatment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xenograft and Collagen membrane (Active Comparator): Placing the implant with collagen membrane and xenograft at esthetic zone of maxillary ridge when 2-4 mm of implant threads exposure .
  Interventions: Procedure: Xenograft and Collagen membrane
- Xenograft and A-PRF (Experimental): Placing the implant with xenograft and A-PRF at esthetic zone of maxillary ridge when 2-4 mm of implant threads exposure .
  Interventions: Procedure: Xenograft and APRF

INTERVENTIONS:
Procedure: Xenograft and Collagen membrane — Placing the implant with collagen membrane and xenograft at esthetic zone of maxillary ridge with 2-4 mm thread exposure .
  Arms: Xenograft and Collagen membrane
Procedure: Xenograft and APRF — Placing the implant with APRF and xenograft at esthetic zone of maxillary ridge with 2-4 mm thread exposure .
  Arms: Xenograft and A-PRF

SUMMARY:
Comparative study for evaluation of vertical bone gain after one stage ridge augmentation with advanced platelet rich fibrin (A-PRF) and xenograft versus guided bone regeneration using collagen membrane and xenograft.

DETAILED DESCRIPTION:
Summry description

* Dental implants represent a reliable mean for replacing missing teeth and restoring dental function.
* With increased use of dental implants in replacement of missing teeth in partially edentulous patients the need for implants that satisfy both esthetics and function .
* Thus, the concept of restoration-driven implant placement has been introduced to provide a good match between the position of implant and the future position of the implant supported-restoration to provide a good clinical outcome.
* The concept of prosthetic-driven implant dimensional changes are expected in the hard and soft tissues.
* About 50% of alveolar bone loss occurs in the buccolingual direction in the first 12 months after tooth extraction.
* The alveolar process can be too narrow to facilitate a complete bony surrounding of the placed dental implant.
* Which may lead to a peri-implant bony dehiscence when placing an implant.
* One stage ridge augmentation procedure has been advocated in management of buccal dehiscence and fenestration defects that may develop with implant placement according to prosthetic-driven implant placement concept.
* Guided bone regeneration techniques (GBR) are commonly used in management of these defects.
* However, controversy still exists concerning the complications that may arise such as membrane exposure and its effects on bone regeneration and the possibility of using bone grafts alone to overcome these problems.
* This research promotes the evaluation of A-PRF in combination with xenograft in one stage ridge augmentation.
* The addition of A-PRF to bone grafts has been reported to enhance the process of bone regeneration through different mechanisms.
* Ridge augmentation according to the principle of GBR using collagen membrane and bone graft has been proven to be predictable in producing significant bone gain promoting implant placement.
* The aim of the study is to clinically evaluate vertical bone gain in buccal peri-implant dehiscence and fenestration defects following application of advanced PRF plus xenograft compared to guided bone regeneration using collagen membrane and xenograft.

Surgical procedure:

- Control group: (Implant placement with xenograft and collagen membrane) After Para crestal incision and raising the mucoperiosteal flap at the top of the alveolar process, the exact position of the dental implant will be defined as determined by preoperative measurements, dental setup, and surgical guide. Bone level implants will be placed 3 mm apical to the expected cervical border of the crown.

The titanium surface of the dental implant will be covered with bone graft (xenograft), and coverage with a resorbable collagen membrane.

-Test group: (implant placement with xenograft and A-PRF) The alveolar bone exposure and implant osteotomy will be prepared and inserted in same manner as in the control group. The titanium surface of the dental implant will be covered with A-PRF and xenograft.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Systemically healthy.
* Has good dental health.
* Missing a single tooth in the maxillary anterior and premolar region
* Crestal residual ridge width of 4-5mm.
* Residual ridge with an adequate band of keratinized tissue (2 mm).
* Residual ridge with sufficient vertical bone height to safely place a >10 mm long dental implant.

Exclusion Criteria:

* Severe parafunctional habits, for example, bruxing and clenching.
* Conditions that complicate wound healing, for example, uncontrolled diabetes (defined as HBA1c level >7%) or smoking.
* Conditions that might lead to a possibly lowered regenerative capacity of the bone, for example, osteoporosis and Paget's disease.
* Pregnant or expecting to be pregnant.
* History of drug and alcohol abuse or certain medications like bisphosphonates or steroids currently or within the past three months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
vertical buccal bone gain | 6 months
  It will be measured using UNC Periodontal probe

SECONDARY OUTCOMES:
horizontal bone gain | 6 months
  It will be measured using UNC Periodontal probe
Ridge width | 6 months
  It will be measured using bone caliper
Post-surgical patient satisfaction | 9 months
  It will be measured using Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah M Shbair, B.D.S, Principal Investigator — Dr
Locations (1):
- Faculty of Dentistry , Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No